CLINICAL TRIAL: NCT00845442
Title: Dynamic Vocal Fold Abduction for Bilateral Paralysis
Brief Title: Dynamic Laryngeal Opening for Bilateral Vocal Fold Paralysis by an Implanted Stimulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 08-03-16; NIH DC-0066854-01; IDE G980179 (Other: Federal Drug Administration)
Record Dates: First submitted 2007-12-26; First posted 2009-02-18 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Vocal Cord Paralysis
Keywords: Bilateral vocal cord paralyses; Implanted laryngeal stimulator; vocal cord opening; pulmonary function tests
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pacemaker — Placement of pacemaker over the chest wall to stimulate the larynx in the neck via a tunneled electrode

SUMMARY:
People who had paralysis of the vocal cords are often prevented from breathing by this problem because the cords will not open, and the patients have to wear a tracheostomy (neck breathing tube) to bypass this airway obstruction. This study examines the effects of vocal cord opening triggered by a pacemaker implanted over the chest wall. The device is connected to a nerve taken from a muscle close to the larynx (voice box) and implanted into the paralysed laryngeal muscle so it can reinnervate it. When this process is complete after a few weeks, the stimulator is turned on and the level of vocal cord opening is assessed. Airway improvement is checked by pulmonary function tests and measurements of vocal cord opening. The ultimate goal of the study is to lead to situations where patients with bilateral vocal fold paralyses could get rid of the neck breathing tube to have less complications, be more comfortable and socially acceptable.

DETAILED DESCRIPTION:
Data pending

ELIGIBILITY:
Inclusion Criteria:

* Breathing difficulties from vocal cord paralyses
* Tracheostomy tube
* Ability to understand the purpose of the research
* Appropriate hand motor coordination

Exclusion Criteria:

* Lack of understanding the research
* Poor hand motor coordination
* Non-acceptance of tracheostomy
* Inability to passively move the paralyzed vocal cords

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2010-11-01 (Actual)

SECONDARY OUTCOMES:
Tolerance of implanted device | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Broniatowski, MD, Principal Investigator — University Hospitals Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States